CLINICAL TRIAL: NCT06926634
Title: Zanzalintinib Maintenance in Patients With High Grade Neuroendocrine Neoplasms (HG-NENs)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202506139
Record Dates: First submitted 2025-04-10; First posted 2025-04-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: High Grade Neuroendocrine Neoplasms
Keywords: High grade; Neuroendocrine tumors; Zanzalintinib; Phase 2
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanzalintinib (Experimental): Zanzalintinib 60 mg taken by mouth once daily in 28-day cycles for up to 3 years.
  Interventions: Drug: Zanzalintinib

INTERVENTIONS:
Drug: Zanzalintinib — Provided by Exelixis

SUMMARY:
The investigators hypothesize that zanzalintinib maintenance therapy after initial cytotoxic chemotherapy can prolong the progression-free survival (PFS) in patients with high-grade NENs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed high-grade poorly differentiated or well differentiated neuroendocrine tumor (with a Ki-67 of ≥20%), excluding small cell lung cancer (SCLC) and Merkel cell cancer. High-grade includes any neuroendocrine neoplasm with a Ki-67 of >20% or with mitotic count of more than 20 mitoses per high power field or any poorly differentiated neoplasm or any neoplasm lacking these that is deemed high grade by pathology consensus, based on other markers (necrosis or IHC demonstrating p53 or RB mutation). This includes:

  * High-grade well-differentiated neuroendocrine neoplasms
  * Transformed NENs from a lower to a higher grade (patient may have some low grade and some high grade NENs)
  * High-grade neoplasms with significant expression of neuroendocrine markers such as synaptophysin, chromogranin or INSM-1 or unknown origin neoplasms with gene expression signatures consistent with neuroendocrine lineage (as per validated tissue of origin testing, such as CancerType ID, after pathology consensus).
  * Mixed neuroendocrine and non-neuroendocrine neoplasms (MiNEN), including MiNEN per WHO and mixed neoplasms not fulfilling criteria of MiNEN. The neuroendocrine component would need to be a high-grade neuroendocrine tumor as documented by pathology review.
  * Note: For ambiguous cases, will consult with a designated expert pathologist.
* Measurable disease per RECIST 1.1.
* Current or prior somatostatin analogue therapy is allowed if clinically indicated.
* Patients must have received their initial course of chemotherapy and be eligible for a chemotherapy break with the most recent disease imaging assessment showing stable disease (SD) or a partial response (PR) by RECIST 1.1. The imaging showing stable disease or partial response should have occurred either during the chemotherapy or right after discontinuation of the chemotherapy treatment and before any other treatment. Reasons for treatment break can include physician or patient preference, completion of pre-specified treatment cycles, or toxicity. Patients intolerant of chemotherapy may also be eligible for the study, but they must have been treated with at least 2 cycles of chemotherapy and at least one imaging assessment on treatment or right after treatment showing PR or SD per RECIST 1.1. There is no limit for prior lines of non-chemotherapeutic regimens (including targeted agents, immunotherapy or radioligand treatment), but the most recent treatment prior to study initiation must contain chemotherapeutic agents.
* At least 18 years of age.
* ECOG performance status ≤ 2 (Karnofsky ≥ 80%).
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 K/cumm without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection.
  * Platelets ≥ 100 K/cumm without transfusion within 2 weeks prior to screening laboratory sample collection.
  * Hemoglobin ≥ 9.0 g/dL without transfusion within 2 weeks prior to screening laboratory sample collection.
  * International Normalized Ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.2 x IULN.
  * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease, total bilirubin ≤ 3 x IULN).
  * Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 x IULN. For subjects with documented bone metastasis, ALP ≤ 5.0 x IULN.
  * Creatinine ≤ 1.5 x IULN OR calculated creatinine clearance ≥ 40 mL/min by Cockcroft-Gault equation.
  * Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤113.2 mg/mmol) creatinine.
* Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from adverse events (AEs), including immune-related adverse events (irAEs), related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (eg, physiological replacement of corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ Grade 2 hypomagnesemia, ≤ Grade 2 neuropathy are permitted.
* Sexually active fertile subjects and their partners must agree to use highly effective method of contraception during the course of the study and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (eg, condom), is required with use of oral contraceptives. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction through 186 days after the last dose of zanzalintinib for women of childbearing potential (WOCBP) or through 96 days after the last dose of zanzalintinib for men.
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met:

  * permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) OR
  * documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause).
  * Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior treatment with zanzalintinib (XL092) or cabozantinib (XL184).
* Another malignancy that requires active therapy and in the opinion of the Investigator would interfere with monitoring of radiologic assessments of response to Investigational Product, within 2 years before C1D1, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy. Incidentally diagnosed prostate cancer is allowed if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.

  * Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
  * Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before C1D1.
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before C1D1.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before C1D1.
* Receipt of strong or moderate CYP3A4 inhibitors or inducers within 4 half-lives of C1D1. (This includes cimetidine, because of its potential to interfere with CYP3A4 mediated metabolism of zanzalintinib.)
* Use of concomitant medications that are known to prolong the QT interval within 4 half-lives of C1D1.
* Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors) and platelet inhibitors (eg, clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardioprotection (per local applicable guidelines) and low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before C1D1 without clinically significant hemorrhagic complications from the anticoagulation regimen.

    * Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to C1D1, whichever is longer.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to zanzalintinib.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Unstable or deteriorating cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).
    * Uncontrolled hypertension defined as sustained blood pressure (BP) ≥ 140 mm Hg systolic or ≥ 90 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic event within 6 months before C1D1.
    * Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous or non-CVA/TIA arterial thromboembolic events within 3 months before C1D1.

      * Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before C1D1 without clinically significant hemorrhagic complications from the anticoagulation regimen.
      * Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the PI.
    * Prior history of myocarditis.
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI-tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless cause of obstruction is definitively managed and subject is asymptomatic
    * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months before first dose.

      * Note: Complete healing of an intra-abdominal abscess must be confirmed before C1D1.
    * Known gastric or esophageal varices
    * Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 4 weeks
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before C1D1.
* Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
* Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta.

  * Note: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following PI approval.
* Other clinically significant disorders that would preclude safe study participation.

  * Active infection requiring systemic treatment.

    * Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.
  * Known infection with acute or chronic hepatitis B or C
  * Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness except for subjects meeting all of the following criteria: (1) on stable anti-retroviral therapy; (2) CD4+ T cell count ≥ 200/µL; and (3) an undetectable viral load.

    * Note: HIV testing will be performed at screening if and as required by local regulation.
    * Note: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose.
    * Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider.
  * Serious non-healing wound/ulcer/bone fracture.

    * Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  * Malabsorption syndrome.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogeneic stem cell transplant.
* Major surgery (as defined in Appendix G; eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to C1D1. Prior laparoscopic surgeries (eg nephrectomy) within 4 weeks prior to C1D1. Minor surgery (eg, simple excision, tooth extraction) within 5 days before C1D1. Complete wound healing from major or minor surgery must have occurred at least prior to C1D1.

  * Note: Fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 2 weeks per electrocardiogram (ECG) before C1D1.

  * Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Inability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of study entry.
* Other conditions, which in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through completion of follow-up (up to 6 years)
  PFS is defined as the time from the date of initiation of zanzalintinib treatment to progression or death, whichever occurs first. The alive patients without progression are censored at the last follow-up.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through completion of follow-up (up to 6 years)
  ORR) is defined as partial response rate (PRR) + complete response rate (CRR) in patients who receive zanzalintinib
Overall survival (OS) | Through completion of follow-up (up to 6 years)
  OS is defined as the time from the start of zanzalintinib treatment to the date of death, censored at the last follow-up otherwise.
Number of participants with adverse events | From start of treatment through 30 days after last dose of zanzalintinib (estimated to be 37 months)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Trikalinos, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu